CLINICAL TRIAL: NCT04069663
Title: Efficacy of Re-challenge With Immune-checkpoints Inhibitors in Advanced Non-Small-Cell Lung Cancer (NSCLC) Patients: a Retrospective Observational Study
Brief Title: Efficacy of Re-challenge With Immune-Checkpoints Inhibitors in Advanced Non-Small-Cell Lung Cancer Patients: a Retrospective Observational Study
Acronym: RE-CHALLENGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: 38RC19.005
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventional study — Retrospective data analysis

SUMMARY:
This is a multicentre, retrospective, national observational study aiming to describe clinical outcomes of advanced NSCLC patients that performed an ICP re-challenge during their history of disease. The objective of this study is to evaluate the ICP re-challenge efficacy.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICP), including nivolumab, pembrolizumab and atezolizumab, are currently approved by EMA (European Medicines Agency) and ANSM (National Agency for the Safety of Medicines and Health Products) for the treatment of advanced Non-Small-Cell Lung Cancer (NSCLC) in first or second line with different strategies according to the expression of PD-L1. Moreover, durvalumab recently entered the treatment strategy for locally advanced disease in PD-L1 expressing (>1%) patients. Median progression-free survival (PFS) for patients with advanced NSCLC is approximately 3 to 4 months with this kind of drugs and chemotherapy is currently the reference treatment after progression. However, the scientific community is now evaluating the re-challenge strategy. Notably, in patients with metastatic melanoma, different trials have shown the efficacy and the good safety of re-challenge with ipilimumab or a combination of nivolumab and ipilimumab after an initial period of disease control with ipilimumab.

To date, no studies have reported the clinical benefit of ICP re-challenge in patients with advanced NSCLC. The effectiveness and tolerance of the re-challenge strategy with the same or another ICP remains therefore a major issue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NSCLC
* Advanced disease (stage III-IV) according to the TNM 7th /8th edition classification at the beginning of first ICP
* Patients must have received at least two lines of ICP during their history of disease
* Patients with EGFR mutation and/or ALK translocation must have received all specific target agents regularly reimbursed (during the reporting period) prior to the first PCI

Exclusion Criteria:

• Opposition form signed by the living patient or opposition clearly indicated in the deceased patient's medical records

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective, French, multicentre cohort
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 year
  Overall Survival

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
  Progression Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Gobinni, MD, Study Director — University Hospital, Grenoble; Matteo Giaj Levra, pHD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hosipital, Grenoble, La Tronche, Isère, France

IPD SHARING:
Plan to Share IPD: No